CLINICAL TRIAL: NCT03434405
Title: Mindfulness-based Social Cognition Group Training for Persons With Diagnoses of Psychotic Disorders (SocialMind): A Feasibility, Non-randomized Controlled Trial
Brief Title: Mindfulness-based Social Cognition Training for Psychosis (SocialMind): A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGES-Mind Feasibility Study
Record Dates: First submitted 2018-02-02; First posted 2018-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-01

CONDITIONS: Schizophrenia and Disorders With Psychotic Feature; Psychotic Episode
Keywords: schizophrenia; mindfulness; social cognition; SocialMind; AGES-Mind
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Multi-center, open-label, prospective, non-randomized, single-group, clinical trial. The experimental arm will receive TAU (both drug and psychosocial therapy) and mindfulness-based social cognition group training (SocialMind), specifically designed for patients with first episode psychosis by the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SocialMind (Experimental): The experimental arm will receive treatment as usual (both psychotropic treatment and psychosocial treatment) and mindfulness-based social cognition group training (SocialMind), specifically designed for patients with first episode psychosis by the research team. There will be a first phase (intensive intervention) consisting of 8 weekly sessions and a second phase (follow-up sessions) consisting of 4 fortnightly sessions and 5 monthly sessions.
  Interventions: Behavioral: SocialMind; Behavioral: Psychosocial treatment; Drug: Psychotropic treatment

INTERVENTIONS:
Behavioral: SocialMind — SocialMind is a mindfulness-based intervention including elements such as radical acceptance, decentering or meditation-techniques. It is designed to target social cognition, defined as the ability to recognize, understand and benefit from social stimuli.
  Other Names: Mindfulness-based social cognition training; Mindfulness-based social cognition group training; MB-SCT
Behavioral: Psychosocial treatment — Treatment as usual delivered by patient's practitioner
Drug: Psychotropic treatment — Treatment as usual delivered by patient's practitioner

SUMMARY:
The current investigation has been designed to test the feasibility of a mindfulness-based social cognition training (SocialMind) for people with a first episode of psychosis (AGES-Mind Study, NCT03309475). The intervention has been designed by professionals with both formal training and clinical experience in the field of mindfulness and third generation cognitive-behavioral therapies. Main outcomes are recruitment rate, adverse events and treatment adherence, although therapy effects and adjustment to intervention manual are also explored.

DETAILED DESCRIPTION:
Social functioning is impaired among many patients with a first episode of psychosis, who also show a lower ability to recognize, understand and benefit from social stimuli (i.e., deficits in social cognition) than their pairs. Both deficits underlie the general functional impairment found across non-affective psychotic syndromes. Since currently available pharmacological strategies have not proven themselves effective in addressing this matter, new psychotherapeutic approaches should be developed. This research team developed a mindfulness-based social cognition group training (SocialMind) designed for persons who have suffered a first episode of psychosis within five years prior to their enrollment in the study (AGES-Mind Study, NCT03309475). Although there is enough evidence to support the lack of adverse events derived for mindfulness-based interventions specifically designed for psychotic patients (Cramer et al., 2016), many clinicians express their concerns about the beneficial effects of these approaches. Therefore, and in keeping with international health organisms such as United Kingdom's National Health Service (NHS), this team have proposed a feasibility study. The main hypothesis is that the AGES-Mind study can be carried out in terms of achievement of recruitment rate, lack of adverse events and levels of treatment adherence. Secondary hypothesis states that clinicians will adhere to SocialMind manual. Finally, a positive effect of the intervention is expected, both in participants' satisfaction and in some relevant variables, such as functional outcomes, clinical global impression and social cognition.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Diagnosis of psychotic disorder according to DSM-5 and history of more than five years of psychotic symptoms
* CGI-SCH equal or lower than four points ("moderately ill")
* Informed consent given

Exclusion Criteria:

* Intellectual disability plus impaired global functioning prior to disorder onset
* Generalized development disorder
* Substance related disorders (except for nicotine) according to DSM-5

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-02-25 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 0 weeks
  At least 25 participants meeting inclusion criteria

SECONDARY OUTCOMES:
Attrition rate | 8 weeks
  Attrition rate lower than 30% on the experimental arm
Change in Psychiatric Symptoms | 8 weeks
  Psychiatric symptoms are measured by the 90 Symptoms Check List Revised (SCL-90-R) that explores 9 domains of psychopathology and provides 3 general scales. Higher values indicate higher symptomatology within each scale.
Change in dissociative Symptoms | 8 weeks
  Dissociative symptoms are measured by Dissociative Experiences Scale (DES-II), a scale that explores the frequency of several dissociative experiences. There is only one scale. Higher values indicate more dissociative experiences
State anxiety | 8 weeks
  State anxiety within sessions (before and after the training) are measured by the State scale of the State-Trait Anxiety Inventory (STAI-S). Higher values indicate higher anxiety symptoms in one general scale.
Participants' satisfaction | 8 weeks
  Client Satisfaction Questionnaire (CSQ-8) is a self-reported measure of therapy satisfaction. It provides one unique dimension, with higher values indicating more satisfaction with the intervention.
Change in clinical global impression | 8 weeks
  Clinical Global Impression Scale for Schizophrenia (CGI-SCH) measures patients' clinical state and clinical change over time. There are four scales (positive, negative, cognitive and depressive symptoms) and one general scale. Higher values indicate a worst clinical impression.
Change in social functioning | 8 weeks
  Personal and Social Performance Scale (PSP) explores four domains of social functioning (self-care, social relationships, social activities and disruptive and aggressive behavior. There are four specific scales from each domain (range 1-7) and one general scale (range 1-100). Higher values indicate worst functioning within each of the four specific areas, but better general functioning in the general scale.
Change quality of life | 8 weeks
  Quality of life is measured by the instrument designed by the World Health Organization WHOQOL-BREF. There is only one dimension, with higher values indicating worst quality of life.
Change in theory of mind | 8 weeks
  Reduced version of the hinting task measures theory of mind ability through five different stories. The test provides one scale (from 0 to 10 points). Higher values indicate better performance.
Change in emotion recognition | 8 weeks
  The Reading the Mind in the Eyes Test (RMET) measures the ability to recognize different complex emotions on several faces. There is only one dimension. Higher values indicate more emotions correctly recognized (from 0 to 40).
Change in social attribution | 8 weeks
  The Attribution Intentions Hostility Questionnaire (AIHQ) measures people's disposition to interpret different ambiguous situations as hostile or neutral. Two main domains are hostility bias and aggression bias. Higher values indicate stronger biases.
Change in reflective functioning | 8 weeks
  Reflective Functioning Questionnaire (RFQ-8) measures mentalization ability through a set of 8 questions. There is only one dimension (from 0 to 56), with higher values indicating a stronger ability to mentalize.
Change in mindful attention and awareness | 8 weeks
  Mindful Attention and Awareness Scale (MAAS) measures this key aspect of mindful disposition. There is only one dimension (from 0 to 90), with higher values indicating better attention and awareness
Change in neurocognitive status | 8 weeks
  Screening of Cognitive Impairment in Psychiatry for Schizophrenia (SCIP-S) explores five major cognitive domains: immediate verbal learning, delayed verbal learning, working memory, verbal fluency and processing speed. There are five specific domains (each of them provides a different cut-off point) and a general scale (less than 67 points suggests cognitive impairment).

OTHER OUTCOMES:
Clinician's adjustment to treatment protocol | 8 weeks
  Independent raters assess practitioner's adherence to treatment manual after analyzing recorded sessions

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fe Bravo, MD, PhD, Principal Investigator — Instituto para la Investigación Biomédica del Hospital Universitario La Paz [La Paz University Hospital Biomedical Research Institute]
Locations (1):
- La Paz University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cramer H, Lauche R, Haller H, Langhorst J, Dobos G. Mindfulness- and Acceptance-based Interventions for Psychosis: A Systematic Review and Meta-analysis. Glob Adv Health Med. 2016 Jan;5(1):30-43. doi: 10.7453/gahmj.2015.083. Epub 2016 Jan 1. PMID 26937312
- [Derived] Mediavilla R, Munoz-Sanjose A, Rodriguez-Vega B, Bayon C, Lahera G, Palao A, Bravo-Ortiz MF. Mindfulness-Based Social Cognition Training (SocialMind) for People With Psychosis: A Feasibility Trial. Front Psychiatry. 2019 May 2;10:299. doi: 10.3389/fpsyt.2019.00299. eCollection 2019. PMID 31118909
- See also: AGES-Mind in ClinicalTrials.gov — https://clinicaltrials.gov/ct2/show/NCT03309475?term=ages+mind&rank=1